CLINICAL TRIAL: NCT00503464
Title: "Assessing Barriers to American Diabetes Association Guideline Adherence"
Brief Title: "Assessing Barriers to ADA Guideline Adherence"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Other Study IDs: #R03 HS016065-01; PAR-04-041
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-07

CONDITIONS: Diabetes
Keywords: guideline; adherence
MeSH Terms: conditions — Diabetes Mellitus

SUMMARY:
This project involves a comprehensive assessment of barriers to diabetes guidelines adherence across 25 practices in the Crozer-Keystone primary care PBRN. A Barrier Assessment Tool (BAT) will be validated to correlate with provider and practice adherence to diabetes care guidelines. The network is part of the Crozer-Keystone Health System located in Delaware County, Pennsylvania, in the southeast quadrant of the Philadelphia metropolitan region.

DETAILED DESCRIPTION:
Study hypothesis: Questionnaire responses about perceived barriers to implementation of diabetes care recommendations, administered to primary care providers and staff, will be shown to correlate with that provider's and practice's success at implementing care guidelines.

Diabetes care in the U.S. consistently fails to meet recommended quality standards. Barriers impede the translation of evidence-based guidelines into sustainable practice. Few studies have considered multiple barriers, and there is a lack of evidence-based strategy in choosing interventions to overcome barriers. This study involves a comprehensive assessment of practice barriers to diabetes guidelines adherence across a primary care network. The BAT based upon a framework proposed by Cabana, et al (1999) will be validated to correlate with provider and practice adherence to diabetes care guidelines. A Diabetes Flow Sheet implemented in our Network to track adherence to guidelines will be assessed and correlated with measured barriers. This organizational strategy will support an evidence-based approach to quality initiative interventions. The BAT will be administered to practice team members: providers, support staff, and practice managers in our Network of 25 primary care practices. Five hypotheses are tested:

A: The BAT measures perceived barriers to adherence to diabetes guidelines, while showing adequate internal consistency and an identifiable subscale structure.

B: The BAT results inversely correlate with practice and provider adherence to ADA guidelines.

C: BAT scores will inversely correlate with use of the Diabetes Flow Sheet.

D: The BAT scores inversely correlate with clinical outcomes (glycemic and lipid control.)

E: Use of the Diabetes Flow Sheet correlates with higher provider and practice adherence to ADA guidelines.

The BAT would then provide the structure for comprehensive assessment of barriers. Study of the Crozer-Keystone PBRN is a real-world laboratory for research in the translation of evidence into diverse practices. The Network is optimally positioned to implement and study this organizational strategy.

ELIGIBILITY:
Inclusion Criteria:

* Crozer-Keystone Health Network primary care (Internal Medicine and Family Medicine) providers and support staff in the 25 primary care practices.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell A. Kaminski, M.D., M.B.A., Principal Investigator — Crozer-Keystone Health Network
Locations (1):
- Crozer-Keystone Health System Practice-Based Research Network, Upland, Pennsylvania, United States